CLINICAL TRIAL: NCT07379593
Title: Validation of the Clinical Decision Support Systems (CDSS) Developed in the EU Horizon PREPARE Project in the Rehabilitative Treatment of Idiopathic Scoliosis
Acronym: PREPARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Scientifico Italiano Colonna Vertebrale (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PREPARE-pros
Record Dates: First submitted 2026-01-15; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Adolescent Idiopathic Scoliosis (AIS)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clinical Impact of the CDSS (Experimental): The study aims to investigate the potential clinical impact of the CDSS on the prescription of rehabilitative treatment for idiopathic scoliosis (IS). Specifically, it seeks to answer the following question:
  Would clinical decisions regarding the treatment of IS have changed if clinicians had access to the information provided by the CDSS to discuss with the patient?
  Interventions: Other: CDSS simulation
- Impact of the CDSS on clinicians (Other): Focus grous designed to explore the perspectives, experiences, and perceptions of physicians regarding the use of the CDSS in daily clinical practice.
  Interventions: Other: Focus group - clinicians
- Impact of the CDSS on Patients (Other): The main objective is to explore patients' perspectives on the implementation of CDSS. The aim is to understand patients' experiences with CDSS, including their interactions with the system and their perceptions of its usefulness and relevance in the care pathway. The study also seeks to identify factors that influence patients' acceptance and usability of CDSS, such as interface design, clarity of information, and alignment with patients' preferences. Finally, we aim to evaluate the impact of CDSS on patient engagement and their satisfaction with the care experience, including the extent to which CDSS facilitate informed decision-making and communication between patients and healthcare providers.
  Interventions: Other: Focus group - patients

INTERVENTIONS:
Other: CDSS simulation — The intervention planned in this study consists of a simulation, carried out by physicians, of the use of a Clinical Decision Support System (CDSS) designed to support informed decision-making in prescribing rehabilitative treatment for idiopathic scoliosis (IS).
  Physicians will continue their routine clinical practice and will subsequently be exposed to the CDSS results for the same cases they had previously assessed, after a three-month interval (the typical period between a visit and a follow-up). This delay is intended to minimize recall bias and to ensure that exposure to the CDSS does not retrospectively influence their therapeutic decisions, thereby avoiding any interference with their daily clinical activity.
  The study will simulate the integration of the CDSS into the clinicians' routine workflow. The CDSS will be developed based on advanced computational models using artificial intelligence, specifically adapted to the rehabilitation context for IS, and created during the f
  Arms: Clinical Impact of the CDSS
Other: Focus group - clinicians — Focus group aimed at exploring how the implementation of the CDSS has influenced the clinical practice of physicians who previously simulated its integration into their professional activity, as well as their decision-making processes and approaches to patient care.
  Arms: Impact of the CDSS on clinicians
Other: Focus group - patients — Two separate focus groups will be organized: one for patients and one for parents. During the sessions, hypothetical clinical scenarios involving the use of CDSS in their care pathway will be presented. The scenarios will be identical for both groups. Participants will be encouraged to share their opinions, thoughts, and feelings regarding CDSS. Facilitators will guide the discussion, ensuring that all participants have the opportunity to express their views and that diverse perspectives are collected.
  Arms: Impact of the CDSS on Patients

SUMMARY:
The study aims to validate both the predictive capacity and the clinical usability of the Clinical Decision Support System (CDSS) developed within the PREPARE project (European Union Grant Agreement 101080288 PREPARE HORIZON-HLTH-2022-TOOL-12-01) for the management of idiopathic scoliosis (IS). This will be achieved through simulation-based studies.

DETAILED DESCRIPTION:
Study Population:

Three participant groups will be included:

* Patients under 18 years who have undergone rehabilitative treatment for idiopathic scoliosis at ISICO's main center in Milan.
* Parents of the included patients.
* Specialist physicians in rehabilitation involved in scoliosis management at ISICO.

All participants must have adequate cognitive and language abilities to take part in discussions and complete questionnaires.

Sample Size:

Part I: Involves the 8 ISICO physicians performing clinical visits.

The main outcome measure is the variation in treatment decisions before and after exposure to the CDSS.

With α = 0.05, power = 80%, and expected effect size (Cohen's d = 0.3), the minimum required sample size is 175 clinical cases.

Parts II-III (Focus Groups):

6-12 patients

6-12 parents

6-10 physicians These group sizes align with qualitative research standards to ensure thematic saturation.

Safety Evaluation:

Adverse events will be monitored, recorded, and assessed by the Data Safety Monitoring Committee (DSMC).

Statistical and Analytical Plan:

Quantitative analysis will evaluate:

The frequency, nature, and motivations behind changes in treatment plans after using CDSS recommendations.

Correlations between CDSS suggestions and clinicians' treatment decisions.

Qualitative analysis will interpret data from focus group discussions to identify patterns, trends, and associations between CDSS recommendations, clinical choices, and possible alternative decisions had the CDSS been applied.

ELIGIBILITY:
Inclusion criteria:

Initial visits or follow-up appointments of patients with IS attending the Milan site of ISICO - Italian Scientific Spine Institute for rehabilitative treatment;

Age between 10 and 18 years;

Informed consent to participate in the study

Exclusion criteria:

Visits not related to the treatment of IS (other spinal conditions);

Patients undergoing treatment at other clinics or hospitals.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Changes in clinical decision | Throughout study completion, an avarage of 6 months
  To assess the impact of the CDSS on clinical decisions, a mixed-methods approach, combining quantitative and qualitative analyses, will be adopted. The primary quantitative outcome measure will be the proportion of clinical cases in which the therapeutic decision changes after exposure to the CDSS, defined as a binary outcome (change vs. no change in treatment plan). Therapeutic decisions made before and after CDSS consultation will be compared within the same case.
  Differences in paired pre- and post-CDSS therapeutic decisions will be evaluated using McNemar's test, which is appropriate for assessing changes in paired binary outcomes. Qualitative analyses will explore clinicians' rationale for decision changes and their perceptions of CDSS influence.

CONTACTS AND LOCATIONS:
Locations (1):
- ISICO - Italian Scientific Spine Institute, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
Aninymized data will be uploaded on a public repository